CLINICAL TRIAL: NCT04930562
Title: A Phase 2, Multicenter Study to Evaluate the Efficacy and Safety of BN101 in Subject With Chronic Graft Versus Host Disease (cGVHD) After at Least Fist Line of Systemic Therapy
Brief Title: Efficacy and Safety of BN101 in Subjects With Chronic Graft Versus Host Disease (cGVHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNova Pharmaceuticals (Shanghai) LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN101-201
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Results first posted 2023-11-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: GVHD, Chronic
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; KD025

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 200mg qd (Experimental): 200mg qd po.
  Interventions: Drug: BN101

INTERVENTIONS:
Drug: BN101 — BN101 is an orally ROCK2 selective inhibitor
  Other Names: belumosudil; KD025

SUMMARY:
This is a phase 2, open-label, multicenter trial to evaluate the efficacy and safety of BN101 in subjects with Chronic Graft Versus Host Disease (cGVHD) after at least First Line of systemic therapy.

DETAILED DESCRIPTION:
Approximately 30 subjects will be enrolled to receive orally administered BN101 200 mg QD (once daily)

Study drug will be administered in 28-day cycles until disease progression or unacceptable toxicity. Subjects may receive study drug in the inpatient or outpatient setting.

Curative Effect analysis The efficacy was analyzed based on MITT The point estimate and 95%CI of ORR were calculated based on the exact probability method of binomial distribution.If applicable, a logistic regression model will be used for multivariate analysis.

Descriptive statistical analyses were provided for all secondary efficacy endpoints.

The following subgroups will be analysed:

* Severe cGVHD (Yes/No)
* Number of organs involved (<4 vs. ≥4)
* Number of previous systemic cGVHD treatment (1 vs. ≥2)
* Duration of cGVHD before inclusion (i.e., from the time of cGVHD diagnosis to the time of inclusion)
* Lung Involvement (Yes/No)

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects at least 18 years of age who have had allogenic hematopoietic cell transplant (HCT).
* Previously received at least 1 and not more than 5 lines of systemic therapy for cGVHD
* Receiving glucocorticoid therapy with a stable dose over the 2 weeks prior to screening;
* Have persistent cGVHD manifestations and systemic therapy is indicated

Exclusion Criteria:

* Subject has not been on a stable dose / regimen of systemic cGVHD treatments for at least 2 weeks prior to screening. (Note: Concomitant corticosteroids, calcineurin inhibitors, sirolimus, MMF, methotrexate, rituximab, and extracorporeal photophoresis (ECP) are acceptable. Systemic investigational GVHD treatments are not permitted).
* Histological relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
* Current treatment with ibrutinib. Prior treatment with ibrutinib is allowed with a washout of at least 28 days prior to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, Prof, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (7):
- China (7):
  - Peking University People's Hospital, Beijing
  - Xinqiao Hospital, Army Medical University, Chongqing
  - Guangzhou First People's Hospital, Guangzhou
  - Nanfang Hospital, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou

REFERENCES:
- [Derived] Wang Y, Wu D, Zhang X, Li Y, He Y, Liu Q, Xuan L, Li Z, Qi K, Sun Y, Wang S, Mo W, Gao L, Hua Y, Wang Y, Zhang Y. A phase II study of belumosudil for chronic graft-versus-host disease in patients who failed at least one line of systemic therapy in China. BMC Med. 2024 Mar 26;22(1):142. doi: 10.1186/s12916-024-03348-5. PMID 38532458

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 200mg qd
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 29
  Other | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 19.78 (3.459)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: OR was defined as the percentage of participants with complete response (CR) or partial response (PR). The OR determination of chronic graft versus host disease (cGVHD) was based on cGVHD response assessment performed by clinicians as per the 2014 National Institutes of Health (NIH) Consensus Development Project for Clinical Trials in cGVHD criteria. CR was defined as the resolution of all manifestations in each organ or site. PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site; and cGVHD progression was defined as the clinically meaningful worsening in 1 or more organs regardless of improvement in other organs.
Time Frame: 12 Months
Population: Analysis was performed on mITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
percentage of participants | 73.3 [54.1 to 87.7]

2. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time (in weeks) from first documentation of response to the time of first documentation of deterioration from best response (e.g., CR to PR, or PR to LR). LOR included the response status of unchanged (LOR-U), mixed (LOR-M), or progression (LOR-P). Per the 2014 NIH Consensus Development Project for Clinical Trials in cGVHD criteria; CR was defined as the resolution of all manifestations in each organ or site; PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site; LOR-M was defined as CR or PR in at least one organ accompanied by progression in another organ, LOR-U was defined as outcomes that did not meet the criteria for CR, PR, progression or mixed response, LOR-P was defined as progression in at least one organ or site without a response in any other organ or site. Kaplan-Meier was used for the analysis.
Time Frame: 12 Months
Population: Analysis was performed on responder population which included participants who received at least 1 dose of study medication and achieved a PR or CR response at any post-baseline response assessment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 200mg qd
Number analyzed (Participants) | 22
weeks | 20.2 [9.71 to NA] — 95% CI upper limit was not available because of the less number of participants with event.

3. Secondary Outcome: Time-to-Response (TTR)
Description: Time-to-response was measured as the time (in weeks) from first dose of study drug to the time of first documentation of response. Response was defined as the participants achieving a PR or CR at any post-baseline response assessment. Per the 2014 NIH Consensus Development Project for Clinical Trials in cGVHD criteria; CR was defined as the resolution of all manifestations in each organ or site and PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site
Time Frame: 12 months
Population: Analysis was performed on responder population.
Measure: Median (Full Range); unit: weeks
Arm/Group | 200mg qd
Number analyzed (Participants) | 22
weeks | 4.29 [3.9 to 48.1]

4. Secondary Outcome: Number of Participants With Best Response in Each Individual Organ
Description: Best response was defined as the percentage of participants with CR or PR. Response was assessed per the 2014 NIH Consensus Development Project for Clinical Trials in cGVHD criteria; CR was defined as the resolution of all manifestations in each organ or site; PR was defined as the improvement in at least 1 organ or site without progression in any other organ or site. Organ response assessment was performed on 9 individual organs: skin, eyes, mouth, esophagus, upper gastrointestinal (GI), lower GI, liver, lungs, and joints and fascia and is reported in this outcome measure.
Time Frame: 12 months
Population: Participants received belumosudil 200 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first. The number of participants analyzed is the number of patients with abnormalities in each organ.
Measure: Number; unit: participants
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
participants
  Skin: number analyzed (Participants) | 20
  Skin | 8
  Eyes: number analyzed (Participants) | 22
  Eyes | 6
  Mouth: number analyzed (Participants) | 22
  Mouth | 12
  Esophagus: number analyzed (Participants) | 5
  Esophagus | 3
  Upper GI tract: number analyzed (Participants) | 3
  Upper GI tract | 2
  Lower GI tract: number analyzed (Participants) | 0
  Liver: number analyzed (Participants) | 9
  Liver | 6
  Lungs: number analyzed (Participants) | 13
  Lungs | 2
  Joints and Fascia: number analyzed (Participants) | 9
  Joints and Fascia | 7

5. Secondary Outcome: Number of Participants With Change From Baseline in Overall Score on Lee cGvHD Symptom Scale at Specified Time Points
Description: Lee cGVHD symptom scale, a patient-reported symptom scale used to measure symptom burden and has 7 subscales (Skin, Eyes and Mouth, Breathing, Eating and Digestion, Muscles and Joints, Energy, and Mental and Emotional) with ratings as follows: 0-Not at all, 1-Slightly, 2-Moderately, 3-Quite a bit, 4-Extremely, with lower values representing better outcome. Score for each subscale was normalized to a score ranged from 0 to 100, where higher score=worse symptoms. An overall Lee cGvHD score was calculated as average of these 7 subscales and it ranged from 0 to 100, where a higher score = worse symptoms. EOT visit was performed within 3 days after the participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication.
Time Frame: Baseline and 12 months
Population: Analysis was performed on mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
Participants
  Total score decline of 7 or more points from baseline | 15
  Total score declined by 7 or more points from baseline on two consecutive assessments | 10

6. Secondary Outcome: Failure-free Survival (FFS)
Description: Failure-free survival was defined as the time (in months) from first dose of study drug to either the start of another new systemic treatment for cGVHD, relapse of the underlying disease or death. If no such events happened, FFS was censored by last response assessment or long term follow up assessment, whichever was the latest and available. Kaplan-Meier survival method was used for the analysis.
Time Frame: 12 months
Population: Participants received belumosudil 200 mg orally QD in each 28-day treatment cycle until disease progression, unacceptable toxicity, or death whichever occurred first
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
months | NA [7.79 to NA] — Median FFS has not yet been reached because there are not sufficient number of participants to start a new systemic treatment for cGVHD, relapse of the underlying disease or death.

7. Secondary Outcome: Time to Next Therapy (TTNT)
Description: The TTNT was defined as the time (in months) from first treatment to the time of new systemic cGVHD treatment. TTNT was censored by last response assessment or long term follow up assessment, whichever was earlier. Kaplan-Meier survival method was used for the analysis.
Time Frame: 12months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
months | NA [8.9 to NA] — Median TTNT has not yet been reached due to an insufficient number of participants with new systemic cGVHD treatment.

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time (in months) from first dose of study drug to the death due to any reason. If there was no death, OS was censored by last visit, last long-term follow-up, or study cut-off date, whichever occurred first. Kaplan-Meier survival method was used for the analysis.
Time Frame: 12months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
months | NA [NA to NA] — Median OS has not yet been reached due to an insufficient number of participants death.

9. Secondary Outcome: Change From Baseline in Corticosteroids Dose
Description: Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. EOT visit was performed within 7 days after the participant's last dose of study drug.
Time Frame: 12months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milligrams per kilogram per day
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
milligrams per kilogram per day | 0.277 (0.202)

10. Secondary Outcome: Number of Participants With Change From Baseline in Calcineurin Inhibitor (CNI) Usage.
Description: Calcineurin inhibitors included systemic tacrolimus and cyclosporine. Number of participants who took CNI at Baseline and had reduction and discontinuation in CNI use as compared to Baseline during the study are reported in this outcome measure. EOT visit was performed within 7 days after the participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication.
Time Frame: 12months
Population: Number of participants who took CNI at Baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | 200mg qd
Number analyzed (Participants) | 20
Participants
  Participants with reduction in CNI dose | 7
  Participants who discontinued CNI | 3

11. Secondary Outcome: Change From Baseline in in Global Severity Rating (GSR) Score by Clinician-reported cGVHD Assessment
Description: The GSR assessment was performed by asking the participants to rate their disease severity of cGVHD symptoms on a 0 to 10-point numeric rating scale, where score 0 indicated 'not at all severe cGVHD symptoms' and score 10 indicated 'most severe cGVHD symptoms possible'. The response was defined using scores from 9 organs: skin, eyes, mouth, esophagus, upper gastrointestinal (GI) track, lower GI tract, liver, lungs, and joints and fascia plus GSR. End of treatment (EOT) visit was performed within 7 days after participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. Change from Baseline was calculated as GSR score at Baseline minus the lowest GSR score on scheduled visits with possible ranges from -10 to 10. The higher the number means the better improvement in cGVHD symptoms. Only those categories in which at least 1 participant had data were reported.
Time Frame: 12months
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
score | 5.4 (1.99)

12. Secondary Outcome: Change From Baseline in Symptom Activity by cGVHD Activity Assessment Participant Self-Report
Description: cGVHD symptom severity was self-reported by participants. Participants were asked to rate their disease symptom severity over the last week on the following questions: skin itching at its worst, moth dryness at its worst, mouth pain at its worst, mouth sensitivity at its worst, main compliant on eyes, symptom severity on eyes. Severity rating was done on a 0 to 10-point numeric rating scare, where score 0 indicated 'not at all severe cGVHD symptoms' and score 10 indicated 'most severe cGVHD symptoms possible'. EOT visit was performed within 7 days after participant's last dose of study drug. Baseline value was defined as valid and last non-missing value obtained within 28 days prior to participant receiving first study medication. Change from Baseline was calculated as the symptom severity score at Baseline minus the lowest symptom severity score on scheduled visits minuswith possible ranges from -10 to 10. The higher the number means the better improvement in cGVHD symptoms.
Time Frame: 12months
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | 200mg qd
Number analyzed (Participants) | 30
score | 2.8 (3.07)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | 200mg qd
All-Cause Mortality (participants affected / at risk) | 5/30
Serious Adverse Events (participants affected / at risk) | 11/30
Other Adverse Events (participants affected / at risk) | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 200mg qd (N=30)
Pneumonia (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Oral infections (Infections and infestations) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Myocarditis (Cardiac disorders) | 1
White blood cell count decreased (Investigations) | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin bacterial infection (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Platelet count decreased (Investigations) | 1
Myasthenia gravis (Nervous system disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 200mg qd (N=30)
Upper respiratory tract infection (Infections and infestations) | 12
Sinus tachycardia (Cardiac disorders) | 11
Pneumonia (Infections and infestations) | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 5
Liver injury (Hepatobiliary disorders) | 5
Hypertension (Blood and lymphatic system disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Blood glucose increased (Investigations) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Respiratory tract infection (Infections and infestations) | 3
Otitis media (Infections and infestations) | 2
Oral infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Gastroenteritis (Gastrointestinal disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Renal injury (Renal and urinary disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Weight decreased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood pressure increased (Investigations) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
headache (Nervous system disorders) | 2
Pyrexia (General disorders) | 2
Influenza like illness (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT04930562/Prot_002.pdf
  • Statistical Analysis Plan (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT04930562/SAP_001.pdf